CLINICAL TRIAL: NCT00428129
Title: An Open Label Clinical Trial of Microplasmin Administered Via the Trellis-8 Infusion System for the Treatment of Acute Iliofemoral Deep Vein Thrombosis
Brief Title: Microplasmin Administered Via the Trellis-8 Infusion System for Treatment of Acute Iliofemoral DVT
Acronym: MAX-DVT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to not pursue uPLi for vascular conditions including DVT.
Sponsor: ThromboGenics (Industry)
Collaborators: Bacchus Vascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-M-005
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Deep Vein Thrombosis
Keywords: Acute Iliofemoral Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — microplasmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: microplasmin

INTERVENTIONS:
Drug: microplasmin — 20mg with Trellis-8 15cm Treatment length 40mg with Trellis-8 30cm Treatment length

SUMMARY:
A single centre, single-arm study to evaluate safety and efficacy of microplasmin administration via the Trellis-8 Infusion System in patients with acute iliofemoral DVT

ELIGIBILITY:
Inclusion Criteria include:

* Patients with radiographically-confirmed acute proximal DVT

Exclusion Criteria include:

* Isolated calf or popliteal vein DVT, based on duplex ultrasound
* Thrombus involving the inferior vena cava (IVC)
* Proximal (e.g. cranial) aspect of thrombus cannot be adequately assessed to level of the iliac veins or inferior vena cava, based on duplex ultrasound.
* Cannot traverse the target vessel segment with guidewire
* Symptomatic pulmonary embolism is present at time of presentation
* Documented history of prior DVT in target extremity
* History of anticoagulants administered for > 30 days for undocumented/ unclear reason (e.g. for reasons other than presence of mechanical cardiac valve, atrial fibrillation, etc.)
* Documented history of thrombophilic disorder, with diagnosis established via previous objective testing (e.g. familial screening for thrombophilia).
* Cannot receive standard secondary prevention pharmacotherapy [i.e. heparin or LMWH and vitamin K antagonists (VKA)] due to contraindications to anticoagulation [e.g. known bleeding diathesis, thrombocytopenia (platelets < 100,000 mm3), heparin induced thrombocytopenia (HIT), known allergy to heparin or warfarin]
* Absolute contraindication to thrombolytic therapy
* Previous central nervous system haemorrhage
* Life expectancy less than 1 year, due to other comorbid condition.
* Previous intervention in target limb to address venous thrombus.
* Target limb has chronic venous insufficiency of C4 or greater severity
* Acute or chronic symptomatic musculoskeletal condition in target limb (e.g. trauma, fracture, severe arthritis).
* Documented patent foramen ovale or other right-to-left cardiac shunt.
* Absolute contraindication to contrast media or renal insufficiency (baseline creatinine >2.0 mg/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Treatment success - treated segment has < 25% residual thrombus AND flow is present following administration of microplasmin | During intervention procedure

SECONDARY OUTCOMES:
Grade of lysis | Upon completion of procedure
Limb patency | Baseline, 48h post procedure, Day-7 and Day-30
Target limb reintervention | Day-7 and Day-30
Clinical outcomes | Baseline, 48h post procedure, Day-7 and Day-30

CONTACTS AND LOCATIONS:
Overall Officials: Gerard O'Sullivan, MD, Principal Investigator — Section of Interventional Radiology, Department of Radiology, University College Hospital, Newcastle Road, Galway
Locations (1):
- Section of Interventional Radiology, Department of Radiology, University College Hospital, Newcastle Road, Galway, Co Galway, Ireland